CLINICAL TRIAL: NCT03494322
Title: EACH: A Randomised Phase II Study Evaluating the Safety and Anti-tumour Activity of the Combination of Avelumab and Cetuximab Relative to Avelumab Monotherapy in Recurrent/Metastatic Head and Neck Squamous Cell Cancer
Brief Title: EACH: Evaluating Avelumab in Combination With Cetuximab in Head and Neck Cancer
Acronym: EACH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/17/0560
Record Dates: First submitted 2018-03-20; First posted 2018-04-11 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — avelumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Randomised phase II study with safety run in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avelumab + cetuximab (Experimental): Patients will receive treatment in 4-week cycles and treatment may continue for up to 1 year.
  Avelumab + cetuximab combination therapy:
  Cycle 1
  * Day 1: Cetuximab 500* mg/m2 given IV over approx 3 hrs
  * Day 15: Cetuximab 500* mg/m2 given IV over approx 2 hrs + avelumab 10 mg/kg given IV over approx 1 hr
  All other cycles:
  - Days 1 and 15: Cetuximab 500* mg/m2 given IV over approx 2 hrs + avelumab 10 mg/kg given IV over approx 1 hr
  *Cetuximab dose will be dependent on outcome of safety run-in.
  There must be a 60 minute break between the administration of cetuximab and avelumab.
  Interventions: Drug: Avelumab; Drug: Cetuximab
- Avelumab monotherapy (Other): Patients will receive treatment in 4-week cycles and treatment may continue for up to 1 year.
  Avelumab monotherapy will be given as follows:
  All cycles Avelumab 10 mg/kg on days 1 and 15 given IV over approximately 1 hour
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/kg given IV
Drug: Cetuximab — Cetuximab 500* mg/m2 given IV
  *Cetuximab dose will be dependent on outcome of safety run-in.
  Arms: Avelumab + cetuximab

SUMMARY:
Head & neck (H&N) cancer is the eighth most common cancer in the UK. Advanced H&N cancer which has come back after treatment or has spread to other parts of the body is incurable and the average life expectancy of these patients is less than a year. New drugs called immune checkpoint inhibitors work with the patient's own immune system to fight cancer. They are used in the clinic to treat a number of cancers, including H&N cancer. It may be possible to make immune checkpoint inhibitors more effective by combining drugs that work in different ways. In effect, attacking the cancer from different angles. Cetuximab is a well-established drug that works by blocking signals that tell cancer cells to grow and divide into more cells. It also engages with the immune system within the tumour. The trial aims to see if giving cetuximab along with an immune checkpoint inhibitor drug called avelumab is better at treating advanced H&N cancer than giving avelumab on its own.

These two drugs have not been given together before, so to start with, the investigator plans to enrol a small number of patients and give the patients avelumab + cetuximab to make sure the combination is safe at the doses chosen. After this, the investigator plans to enrol 114 patients with advanced H&N cancer. Half the patients will be treated with avelumab alone and the other half with avelumab + cetuximab. Both drugs are given intravenously in the hospital once every 2 weeks.

Treatment lasts for up to a year and patients will be followed up for up to 2 years from the time they enter the study. Patients will be recruited from around 15 hospitals in the UK. Recruitment would be expected to start in the second quarter of 2018 and it will take about 29 months (Safety run-in: 5 months; Phase II: 24 months) to recruit all the patients.

DETAILED DESCRIPTION:
This is a randomised phase II study comparing the efficacy of avelumab alone with avelumab + cetuximab combination in patients with platinum-resistant advanced or metastatic head & neck cancer. The randomised phase II part of the trial will be preceded by a safety run-in.The objective of the safety run in is to make sure the combination of cetuximab and avelumab at the doses selected for the study are safe and tolerable.

In phase II, the main question the investigator wants to answer is whether or not giving avelumab and cetuximab together is better than giving avelumab alone to treat patients with head and neck cancer that have had previous treatment with cisplatin and whose cancer has come back or spread to other parts of the body. The investigator will compare the number of patients in each group whose cancer has not gotten any worse 6 months after joining the study.

The phase II part of the trial will recruit patients with head & neck squamous cell carcinoma only. However, during the safety run-in, patients with other types of squamous cell carcinomas will also be eligible.

Target accrual:

Safety run-in: up to 16 patients with squamous cell carcinomas; Phase II: 114 patients with head & neck squamous cell cancer

The safety run-in will recruit patients in cohorts of 3 at a time and all patients will be treated with the combination. The safety run in is a dose de-escalation design. That is, patients will be given the dose that is planed for use in phase II and if this proves not tolerable, the dose of cetuximab will be de-escalated and another cohort of patients will be recruited. The investigator will conclude the combination is safe and tolerable if less than 33% of patients who are treated experience side effects that lead to a dose reduction. The purpose is to ensure the safety of the combination prior to starting phase II, as these drugs have not been given together before. However, there is evidence from previous studies that these types of drugs can be combined safely. The trial aims to complete the safety run-in within 5 months and the phase II study within 24 months. The entire duration of recruitment is expected to be 29 months.

ELIGIBILITY:
Inclusion Criteria:

1. Safety run in: Histologically or cytologically confirmed recurrent or metastatic squamous cell carcinoma that is considered incurable by local therapies

   Phase II: Histologically/cytologically confirmed recurrent/metastatic squamous cell carcinoma of the head and neck that is considered incurable by local therapies.
2. Prior treatment with a platinum agent (either for recurrent/metastatic disease; or as part of radical intent multimodality treatment if disease has recurred within 6 months). (NB: This criterion is not applicable for the safety run-in).
3. No previous treatment with cetuximab for metastatic/recurrent disease
4. Age ≥18 years
5. WHO Performance Status 0 or 1
6. Measurable disease according to RECIST v1.1
7. Adequate bone marrow function
8. Adequate liver function
9. Adequate renal function
10. Adequate venous access for administration of treatment and collection blood samples for exploratory biological samples
11. Willing to have a new biopsy (NB: This criterion is not applicable for the safety run-in).
12. Life expectancy of >3 months
13. Women of child-bearing potential and male patients with partners of child-bearing potential must agree to use adequate contraception methods from date of informed consent, which must be continued for 120 days after completion of trial treatment.
14. Able to give informed consent, indicating that the patient has been informed of and understands the experimental nature of the study, possible risks and benefits, trial procedures, and alternative options
15. Willing and able to comply with the protocol for the duration of the study, including the treatment plan, investigations required and follow up visits.

Exclusion Criteria:

1. Patients with undifferentiated nasopharyngeal or sino-nasal cancers.
2. Disease suitable for treatment with curative intent.
3. Prior therapy with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent.
4. Treatment with any investigational agent within 4 weeks prior to the first dose of trial treatment.
5. Anti-cancer monoclonal antibody therapy within 4 weeks prior to randomisation
6. Chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks prior to randomisation.
7. Persisting grade ≥2 toxicity related to prior therapy
8. Patients with concurrent or previous malignancy that could compromise assessment of the primary or secondary endpoints of the trial.
9. Women who are pregnant or breast feeding.
10. Grade 3 or 4 peripheral neuropathy.
11. Any serious and/or unstable pre-existing medical, psychiatric or other condition, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Patients who are not able to give informed consent for any reason.
13. Active central nervous system (CNS) metastases and/or carcinomatous meningitis
14. Hepatitis infection at screening
15. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
16. Prior organ transplantation including allogenic stem-cell transplantation
17. Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
18. Active infection requiring systemic therapy
19. Has received a live vaccine within 28 days prior to first dose of trial treatment
20. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (n.b. the use of physiologic doses of corticosteroids may be approved after consultation with UCL CTC)
21. Active autoimmune disease that might deteriorate when receiving an immune-stimulatory agent.
22. Current use of immunosuppressive medication
23. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e. bronchiolitis obliterans, cryptogenic organising pneumonia), or evidence of active pneumonitis on screening chest CT scan. (History of radiation pneumonitis in the radiation field is permitted).
24. Significant cardiovascular disease
25. Known prior severe hypersensitivity to either investigational product or any component in their formulations, including known severe hypersensitivity reactions to monoclonal antibodies
26. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis.
27. Patients with a history of keratitis, ulcerative keratitis or severe dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety run-in: Occurrence of dose limiting toxicity | From start of cycle 1 (each cycle is 28 days) upto six weeks.
  Detailed adverse event monitoring will be conducted according to CTCAE v4.03. Patients experiencing any of the following adverse events related to either cetuximab or avelumab during the DLT period will be considered to have experienced a DLT:
  * Any grade 3 or 4 adverse reaction requiring a dose reduction of cetuximab
  * Any adverse reaction resulting in a more than a 14 day treatment delay for any agent.
Phase II: Disease control rate at 24 weeks after randomisation | From randomisation upto 24 weeks
  Assessed using iRECIST

SECONDARY OUTCOMES:
Objective response (iCR or iPR) at 6 and 12 months | 6 months and 12 months after registration/randomisation
  Using iRECIST
Disease control at 6 and 12 months | 6 and 12 months after registration/randomisation
  Using iRECIST
Best overall response | From start of treatment to 24 months after registration, or upto start date of a new treatment for their disease, whichever came first, assessed up to 24 months.
  Using iRECIST
Duration of response | From the date of the first response assessment showing iCR or iPR to the date of the response assessment documenting iPD according to iRECIST, assessed up to 24 months.
  Using iRECIST
Overall survival | Time from registration/randomisation to death from any cause, assessed up to 24 months.
Time to Progression | From date of registration/randomisation to date of first documented progression, assessed up to 24 months.
Progression free survival | From date of registration/ randomisation to date of first documented progression, assessed up to 24 months.
Frequency and severity of adverse events | From informed consent to 90 days post last IMP treatment
Treatment related dose delays or treatment discontinuation | From start of treatment to end of treatment, assessed up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, FRCP PhD, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Ng K, Metcalf R, Sacco J, Kong A, Wheeler G, Forsyth S, Bhat R, Ward J, Ensell L, Lowe H, Spanswick V, Hartley J, White L, Lloyd-Dehler E, Forster M. Protocol for the EACH trial: a multicentre phase II study evaluating the safety and antitumour activity of the combination of avelumab, an anti-PD-L1 agent, and cetuximab, as any line treatment for patients with recurrent/metastatic head and neck squamous cell cancer (HNSCC) in the UK. BMJ Open. 2023 Nov 27;13(11):e070391. doi: 10.1136/bmjopen-2022-070391. PMID 38011968